CLINICAL TRIAL: NCT05151263
Title: Prevalence of Aspirin Resistance in Ischemic Stroke Patients at Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Saeed Mostafa, principal investigator, Assiut University
Other Study IDs: aspirin resistance in stroke
Record Dates: First submitted 2021-11-28; First posted 2021-12-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Acetyl Salicylate — Aspirin is an effective antiplatelet agent, exhibiting its action by irreversibly inhibiting platelet cyclooxygenase-1 enzyme, thus preventing the production of thromboxane A2 (TXA2). It has been used in the primary and secondary prevention of thromboembolic vascular events
  Other Names: aspirin
Diagnostic Test: Optical Platelet Aggregation test — The evaluation of platelet aggregation was performed using an optical aggregometer (AggRAM, using fresh citrated blood. Platelet-rich plasma was obtained by centrifugation of the citrated blood at 190 g for 5 min. The platelet count was adjusted to 200,000 to 300,000 platelets/mm3. Platelet-rich plasma (250 μl) was deposited in each equipment channel, and the activators adenosine diphosphate, epinephrine, collagen, and arachidonic acid were used according to the manufacturer's instructions. aspirin resistance was defined as platelet aggregation ≥ 20% with arachidonic acid and ≥70% with adenosine diphosphate.

SUMMARY:
* This study aims to assess the prevalence of aspirin resistance in patients with acute ischemic stroke and its importance in secondary stroke prevention.
* Effect of aspirin resistance on short and long term mortality and detection of its relationship with recurrence of stroke.

DETAILED DESCRIPTION:
Stroke is the rapidly developing loss of brain functions due to disturbance in the blood supply to the brain. It is the leading cause of adult disability in the United States and Europe and currently the second leading cause of death, ranking after heart disease and before cancer, accounting for 10% of deaths worldwide . About 80-90% of strokes are caused by ischemia, and the remainder by hemorrhage . Arterioarterial micro thromboembolism is an important etiological factor in the pathogenesis of ischemic stroke. Platelet activation in cerebrovascular disease is associated with recurrent stroke and death, while inhibition of platelet function by antiplatelet drugs including aspirin lowers the risk of ischemic stroke. Aspirin is an effective antiplatelet agent, exhibiting its action by irreversibly inhibiting platelet cyclooxygenase-1 enzyme, thus preventing the production of thromboxane A2 (TXA2). It has been used in the primary and secondary prevention of thromboembolic vascular events. Yet, some patients experience recurrent ischemic events despite optimal antiplatelet therapy. This has raised the possibility that these patients may be resistant to aspirin and generated much interest in identification of such patients with laboratory tests of platelet function. Although many studies have demonstrated aspirin resistance in cardiovascular disorders including coronary artery disease, metabolic syndrome , and diabetes by certain tests of aspirin resistance, there are still concerns that these tests have not correlated closely with subsequent recurrent events, and have not reliably identified non-responders to antiplatelet therapy . In addition to the absence of any standardized approach to the diagnosis, there is currently no proven effective treatment for aspirin resistance. Although aspirin resistance has been demonstrated as a possible risk factor for recurrent cardiovascular ischemic events, there is a lack of data correlating aspirin resistance and risk of cerebrovascular ischemic events

ELIGIBILITY:
Inclusion Criteria:

1. At least 7 days of aspirin therapy (acetylsalicylic acid, 100 mg daily) prior to stroke onset
2. Within 24 h of experiencing a new focal or global neurological deficit.
3. Evidence of new or old ischemic infarct on CT brain or magnetic resonance imaging (MRI).
4. With informed consents.
5. Presence or not previous cerebrovascular event as previous history of transient ischemic attack (TIA) before the onset of stroke.

Exclusion Criteria:

1. Patients with other neurological deficits due to stroke mimics or hemorrhagic insult.
2. Patients is subjected to anticoagulant treatment (atrial fibrillation, valve replacement, others).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting consecutively to the Department of Neurology of Assiut university Hospital with acute ischemic stroke whether new onset or recurrent. Acute ischemic stroke was defined as focal neurological deficit persisting for more than 24 h with evidence of cerebral infarction on neuroimaging (MRI brain). The time between stroke occurrence and admission to the hospital was 1-48 h.
Sampling Method: Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
clinical assessment of patients with ischemic stroke | 15-30 min
  assessment of ischemic stroke patient using National Institute of Health Stroke Scale (NIHSS)which is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
  Score Stroke severity 0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
detection of aspirin resistance prevalence between ischemic stroke patients as risk factors and prevention of its recurrence. | 7-10 days
  Prevalence of aspirin resistance between patients of acute new onset stroke are calculated .and among patients with recurrent stroke on aspirin antiplatelet therapy who has aspirin resistance as risk factor calculated. Patients with aspirin resistance shifted to other antiplatelet therapy and MRS (modified Rankin score) evaluated on discharge
clinical assessment of patients with ischemic stroke | 10-15 min
  assessment of ischemic stroke patient using modified Rankin score (MRS).The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bennett D, Yan B, Macgregor L, Eccleston D, Davis SM. A pilot study of resistance to aspirin in stroke patients. J Clin Neurosci. 2008 Nov;15(11):1204-9. doi: 10.1016/j.jocn.2008.01.006. Epub 2008 Sep 27. PMID 18824358
- [Background] Feigin VL. Stroke epidemiology in the developing world. Lancet. 2005 Jun 25-Jul 1;365(9478):2160-1. doi: 10.1016/S0140-6736(05)66755-4. No abstract available. PMID 15978910
- [Background] Donnan GA, Fisher M, Macleod M, Davis SM. Stroke. Lancet. 2008 May 10;371(9624):1612-23. doi: 10.1016/S0140-6736(08)60694-7. PMID 18468545
- [Background] Bogousslavsky J, Van Melle G, Regli F. The Lausanne Stroke Registry: analysis of 1,000 consecutive patients with first stroke. Stroke. 1988 Sep;19(9):1083-92. doi: 10.1161/01.str.19.9.1083. PMID 3413804
- [Background] Yip HK, Liou CW, Chang HW, Lan MY, Liu JS, Chen MC. Link between platelet activity and outcomes after an ischemic stroke. Cerebrovasc Dis. 2005;20(2):120-8. doi: 10.1159/000086802. Epub 2005 Jul 5. PMID 16006760
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Randomised trial of intravenous streptokinase, oral aspirin, both, or neither among 17,187 cases of suspected acute myocardial infarction: ISIS-2. ISIS-2 (Second International Study of Infarct Survival) Collaborative Group. Lancet. 1988 Aug 13;2(8607):349-60. PMID 2899772
- [Background] Zimmermann N, Wenk A, Kim U, Kienzle P, Weber AA, Gams E, Schror K, Hohlfeld T. Functional and biochemical evaluation of platelet aspirin resistance after coronary artery bypass surgery. Circulation. 2003 Aug 5;108(5):542-7. doi: 10.1161/01.CIR.0000081770.51929.5A. Epub 2003 Jul 21. PMID 12874188
- [Background] Borna C, Lazarowski E, van Heusden C, Ohlin H, Erlinge D. Resistance to aspirin is increased by ST-elevation myocardial infarction and correlates with adenosine diphosphate levels. Thromb J. 2005 Jul 26;3:10. doi: 10.1186/1477-9560-3-10. PMID 16045804
- [Background] Kahraman G, Sahin T, Kilic T, Baytugan NZ, Agacdiken A, Ural E, Ural D, Komsuoglu B. The frequency of aspirin resistance and its risk factors in patients with metabolic syndrome. Int J Cardiol. 2007 Feb 14;115(3):391-6. doi: 10.1016/j.ijcard.2006.10.025. Epub 2007 Jan 9. PMID 17218028
- [Background] Watala C, Pluta J, Golanski J, Rozalski M, Czyz M, Trojanowski Z, Drzewoski J. Increased protein glycation in diabetes mellitus is associated with decreased aspirin-mediated protein acetylation and reduced sensitivity of blood platelets to aspirin. J Mol Med (Berl). 2005 Feb;83(2):148-58. doi: 10.1007/s00109-004-0600-x. Epub 2004 Nov 10. PMID 15723265
- [Background] Fateh-Moghadam S, Plockinger U, Cabeza N, Htun P, Reuter T, Ersel S, Gawaz M, Dietz R, Bocksch W. Prevalence of aspirin resistance in patients with type 2 diabetes. Acta Diabetol. 2005 Jun;42(2):99-103. doi: 10.1007/s00592-005-0186-y. PMID 15944844
- [Background] Gorog DA, Sweeny JM, Fuster V. Antiplatelet drug 'resistance'. Part 2: laboratory resistance to antiplatelet drugs-fact or artifact? Nat Rev Cardiol. 2009 May;6(5):365-73. doi: 10.1038/nrcardio.2009.13. Epub 2009 Apr 14. PMID 19365406
- [Background] Lev EI. Aspirin resistance transient laboratory finding or important clinical entity? J Am Coll Cardiol. 2009 Feb 24;53(8):678-80. doi: 10.1016/j.jacc.2008.11.018. No abstract available. PMID 19232900
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950